CLINICAL TRIAL: NCT03953820
Title: Randomized, Open-Label, 2-Way Crossover, 3-Period Study to Evaluate Single Doses of Diazepam Buccal Film Compared With Diazepam Rectal Gel in Adult Males and Females on Concomitant Antiepileptic Drugs for the Treatment of Epilepsy
Brief Title: Diazepam Buccal Film (DBF) - Diastat Rectal Gel (DRG) Crossover Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aquestive Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 180323
Record Dates: First submitted 2019-04-26; First posted 2019-05-17 (Actual); Results first posted 2020-08-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-03

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Diagnosis-Related Groups

STUDY DESIGN:
Intervention Model Description: The study consisted of 2 periods. In Period 1 , participants received a single dose of Diazepam Buccal Film or Diastat Rectal Gel in a randomized sequence following a moderate fat meal with a 28-day washout between doses. Subjects who completed Period 1 were asked to participate in a second period (Period 2) on a voluntary basis. Those subjects who agreed to participate in Period 2 received a second dose of DBF in exactly the same dose and manner as the earlier dose with the exception it was administered following a high fat meal.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Diazepam Buccal Film, Then Diastat Rectal Gel (Experimental): Participants received a single dose of Diazepam Buccal Film following a moderate-fat meal and then received a single dose of Diastat Rectal Gel following a moderate-fat meal with a 28-day washout between doses.
  Interventions: Drug: Diazepam Buccal Film; Drug: Diastat® Rectal Gel (Valeant Pharmaceuticals USA)
- Diastat Rectal Gel, Then Diazepam Buccal Film (Experimental): Participants received a single dose of Diastat Rectal Gel following a moderate-fat meal and then received a single dose of Diazepam Buccal Film following a moderate-fat meal with a 28-day washout between doses.
  Interventions: Drug: Diazepam Buccal Film; Drug: Diastat® Rectal Gel (Valeant Pharmaceuticals USA)
- Diazepam Buccal Film following a High-Fat Meal (Experimental): Participants who volunteered to participate in the second period received a second dose of Diazepam Buccal Film at the same dose and exactly the same manner as the earlier dose with the exception that the dose was administered following ingestion of a high-fat meal.
  Interventions: Drug: Diazepam Buccal Film

INTERVENTIONS:
Drug: Diazepam Buccal Film — Diazepam Buccal Film administered on inner aspect of the cheek at the recommended dose regimen (10 mg to 17.5 mg according to body weight) following ingestion of a moderate fat meal and following ingestion of a high-fat meal.
  Other Names: DBF
Drug: Diastat® Rectal Gel (Valeant Pharmaceuticals USA) — Diastat Rectal Gel administered rectally according to product label administration and dosing instructions (10 mg to 20 mg according to body weight) following ingestion of a moderate-fat meal.
  Other Names: DRG
  Arms: Diastat Rectal Gel, Then Diazepam Buccal Film; Diazepam Buccal Film, Then Diastat Rectal Gel

SUMMARY:
This was a multiple centers, single-dose, open-label, randomized two-sequence crossover, two-period study to evaluate the pharmacokinetics (PK) of single doses of Diazepam Buccal Film (DBF) compared with Diastat® Rectal Gel (DRG) under fed conditions in adult male and female participants on a stable concomitant regimen of anti-epileptic drugs for the treatment of epilepsy.

DETAILED DESCRIPTION:
Period 1 was a randomized, 2-sequence, crossover study in which participants received DBF and DRG following a moderate-fat meal in a randomized sequence with a washout period of 28 days between doses. DBF dose was based on body weight according to the currently recommended dose regimen (derived by Aquestive from population PK modeling in healthy volunteers). DRG dose was based on body weight according to the current product labeling for DRG.

Period 2: Participants who completed Period 1 were asked to participate in a second period on a voluntary basis during which volunteers received a second dose of DBF administered at the same dose and in exactly the same manner as the earlier dose of DBF with the exception that DBF was administered following a high-fat meal.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, smoker (no more than 25 cigarettes or equivalent daily) or non-smoker, ≥ 18 and ≤ 65 years of age, with body weight between 38 and 111 kg, inclusive. Potential subjects with weights in the range of 112 to 134 kg (247 - 249 pounds) may be allowed to participate in the study at the discretion of the Principal Investigator.
2. On a stable and ongoing regimen of at least one AED for treatment of epilepsy. Stable regimen is defined as no change in AED regimen for at least 30 days before the first study drug administration and no change anticipated in the prescribed AED regimen over the course of study participation.
3. Subjects must have a diagnosis of seizure disorder (any seizure type or frequency) under treatment with at least one AED.
4. Healthy (except for seizure disorder), according to the medical history, ECG, vital signs, laboratory results and physical examination as determined by the Principal Investigator/Sub- Investigator.
5. Clinical laboratory values within local laboratories acceptable ranges, unless values are deemed by the Principal Investigator/Sub-Investigator as "Not Clinically Significant".
6. Ability to comprehend and be informed of the nature of the study, as assessed by clinic staff.
7. Availability to volunteer for the entire study duration and willing to adhere to all protocol requirements.
8. Agree not to have a tattoo or tongue or body piercing until the end of the study.
9. Agree not to drive or operate heavy machinery if feeling dizzy or drowsy following drug administration until full mental alertness is regained.
10. Subjects must be able and willing to remove denture or bracing at the time of dosing.
11. Non-vasectomized male subjects must use two forms of medically accepted method of contraception with all sexual partners of childbearing potential during the study and for 111 days following the last dose of study drug. Medically accepted effective forms of contraception include:

    1. simultaneous use of a male condom and
    2. for the female partner, hormonal contraceptives (used since at least 4 weeks) or intrauterine contraceptive device (placed since at least 4 weeks) or diaphragm or cervical cap with intravaginally applied spermicide.
12. Male subjects must be willing not to donate sperm until 111 days following the last study drug administration.
13. Female subjects who are sexually active with a non-sterile male partner (sterile male partners are defined as men vasectomized since at least 6 months) must fulfill at least one of the following:

    1. Be surgically sterile for a minimum of 6 months;
    2. Post-menopausal for a minimum of 1 year;
    3. Agree to avoid pregnancy and use medically acceptable method of contraception as described below until at least 51 days after the last PK blood sample collection of the study. Medically acceptable methods of contraception include:

       * Intrauterine device (hormonal and non-hormonal) placed at least 4 weeks prior to first study drug administration,
       * Oral or transdermal hormonal contraceptives with a 28-days treatment cycle taken daily from at least 30 days prior to first study drug administration and with no expected change in dosage throughout the study, or • Double barrier method (male condom and intravaginally applied spermicide used simultaneously with diaphragm or cervical cap) starting at least 21 days prior to first study drug administration;
    4. agree to complete abstinence.

Exclusion Criteria:

1. Clinically significant abnormal laboratory test results found during medical screening.
2. Positive pregnancy test at screening.
3. Known presence of any clinically significant: hepatic (e.g. hepatic impairment), renal/genitourinary (renal impairment, kidney stones), gastrointestinal (e.g. ulcerative colitis, ileus, partial or complete intestinal blockage, appendicitis), cardiovascular (e.g. uncontrolled hypertension), cerebrovascular, pulmonary, endocrine (controlled diabetes is acceptable), immunological, musculoskeletal, neurological (other than known seizure disorder), psychiatric, dermatological or hematological disease or condition unless determined as not clinically significant by the Principal Investigator/Sub-Investigator and confirmed by Sponsor via written communication prior to subject enrollment.
4. Presence of any clinically significant gastrointestinal pathology (e.g. chronic diarrhea, inflammatory bowel disease), unresolved gastrointestinal symptoms (e.g. diarrhea, vomiting), or other conditions known to interfere with the absorption, distribution, metabolism or excretion of the study drug experienced within 7 days prior to first study drug administration, as determined by the Principal Investigator/Sub-Investigator.
5. Any clinically significant rectal abnormality by history or physical examination, or any condition, for which, in the judgment of the Principal Investigator/Sub-Investigator, administration of rectal gel would cause a potential risk to the subject.
6. Baseline levels of concomitant AED outside of the acceptable therapeutic range at screening.
7. Presence of any clinically significant illness within 30 days prior to first study drug administration, as determined by the Principal Investigator/Sub-Investigator.
8. Presence of any clinically significant physical or organ abnormality as determined by the Principal Investigator/Sub-Investigator.
9. Presence of any clinically significant lesion of the oral cavity.
10. Clinically significant ECG abnormalities (QTcF interval > 450 msec for males or QTcF interval > 470 msec for females) or vital sign abnormalities (systolic blood pressure lower than 90 or over 160 mmHg, diastolic blood pressure lower than 50 or over 100 mmHg, or heart rate less than 50 or over 100 bpm) at screening, unless deemed otherwise by the Principal Investigator/Sub-Investigator.
11. A positive test result for HIV, Hepatitis B surface antigen, Hepatitis C.
12. A positive test result for any of the following: drugs of abuse (amphetamines, methamphetamines, barbiturates, cocaine, opiates, phencyclidine, tetrahydrocannabinol,MDMA, methadone, and benzodiazepines, except where a positive test is consistent with a stable regimen of a prescribed medication) and alcohol breath test.
13. Known history or presence of:

    1. Alcohol abuse or dependence within one year prior to screening;
    2. Drug abuse or dependence;
    3. Hypersensitivity or idiosyncratic reaction to diazepam, DBF excipients, DRG excipients;
    4. Glaucoma (open or acute narrow angle);
    5. Food allergies and/or presence of any dietary restrictions that, in the judgment of the investigator or the Sponsor, would interfere with study procedures or the subject's safe participation in the study.
    6. Severe allergic reactions (e.g. anaphylactic reactions, angioedema).
14. Intolerance to and/or difficulty with blood sampling through venipuncture.
15. Individuals who have donated, in the days prior to first study drug administration:

    * 50-499 mL of blood in the previous 30 days;
    * 500 mL or more in the previous 56 days.
16. Donation of plasma by plasmapheresis within 7 days prior to first study drug administration.
17. Individuals who have participated in another clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to the first dosing, administration of a biological product in the context of a clinical research study within 90 days prior to the first dosing, or concomitant participation in an investigational study including an investigational study involving no drug or device administration.
18. Use of diazepam within 30 days prior to first study drug administration.
19. Use of strong inhibitors of CYP enzymes (e.g. cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem and HIV antivirals) in the previous 30 days before first study drug administration. Use of strong inducers of CYP enzymes (e.g. barbiturates, carbamazepine, glucocorticoids, phenytoin, St. John´s Wort, and rifampicin) and AEDs known to induce CYP enzymes are permitted provided that the regimen of such drugs is stable (taken at least q.d. on a regular basis) within 30 days prior to first study drug administration and until 10 days after last study drug administration.
20. Use of any prescription medication (other than non-systemic topical products) within 30 days prior to first study drug administration. A prescription drug (other than diazepam and any benzodiazepines, phenothiazines, and strong inhibitors of CYP enzymes) that is part of a stable drug regimen (taken at least q.d. on a regular basis) is allowed if taken from at least 30 days prior to the first study drug administration and if there is no expected change in dosage throughout the study.
21. Use of any OTC medications (other than spermicidal/barrier contraceptive products and nonsystemic topical products), within 30 days prior to first study drug administration. OTC drugs that is part of a stable drug regimen (taken at least q.d. on a regular basis) is allowed if taken from at least 30 days prior to the first study drug administration and if there is no expected change in dosage throughout the study.
22. Natural health products (including oral multivitamins, herbal and/or dietary supplements and/or teas) from 30 days pre-dose until after the last PK blood sample collection of each period.
23. Use of marijuana and THC containing products within 3 months prior to screening unless such products are a part of the subject's stable antiepileptic regimen.
24. Use of any monoamine oxidase (MAO) inhibitors (e.g. phenelzine, tranylcypromine), phenothiazines (e.g. chlorpromazine) within 30 days prior to first study drug administration.
25. Female subjects who have taken oral or transdermal hormonal contraceptives (other than 28-days treatment cycle contraceptive products) within 30 days prior to first drug administration, or have used an implanted, injected, or intravaginal contraceptive within 6 months prior to first drug administration.
26. Individuals having undergone any major surgery within 6 months prior to the start of the study, unless deemed otherwise by Principal Investigator/Sub-Investigator.
27. Presence of mouth jewellery, dentures, braces, or piercings in the mouth or tongue that, in the opinion of the Principal Investigator, would be likely to interfere with successful completion of the dosing procedure
28. Dental procedures performed within 14 days of dosing or dental procedures scheduled to occur during study duration.
29. Unable or unwilling to provide informed consent.
30. Have had a tattoo or body/mouth piercing within 30 days prior to first study drug administration.
31. Employee or immediate relative of an employee of Aquestive Therapeutics, any of its affiliates or partners, of the CRO, or the clinical site.
32. Breast-feeding subject.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-04-13 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Slatko, MD, Study Chair — Aquestive Therapeutics
Locations (3):
- United States (3):
  - Clinical Trials of Florida, LLC, Miami, Florida
  - Bioclinica Research, Orlando, Florida
  - Florida Premier Research Institute, LLC, Winter Park, Florida

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 43 healthy (except for seizure disorder) volunteers were screened for eligibility in this study.
Pre-assignment Details: 31 of the 43 screening participants were enrolled and randomized at 5 study sites in the United States. Of those not randomized, 7 did not meet protocol eligibility criteria and 5 were judged eligible but decided not to participate or were not selected to participate in the study since there was already a sufficient number of subjects.
Groups:
- Diazepam Buccal Film, Then Diastat Rectal Gel: Subjects received a single dose of Diazepam Buccal Film and Diastat Rectal Gel following a moderate-fat meal in a randomized sequence with a 28-day washout period between doses.
  Diazepam Buccal Film was administered on the inner aspect of the cheek according to the recommended dose regimen (10 mg to 17.5 mg according to body weight) allowing transbuccal absorption of diazepam.
- Diastat Rectal Gel, Then Diazepam Buccal Film: Subjects received a single dose of Diastat Rectal Gel and Diazepam Buccal Film following a moderate-fat meal in a randomized sequence with a 28-day washout period between doses.
  Diastat Rectal Gel was administered rectally according to package insert dosing instructions (10 mg to 20 mg according to body weight) allowing rectal absorption of diazepam.
- Diazepam Buccal Film Following a High-Fat Meal: Subjects who completed Periods 1 and 2 were asked to participate in Period 3 on a voluntary basis.
  Subjects who volunteered to participate in Period 3 received a second dose of DBF at the same dose and in the same manner as the earlier dose of DBF with the exception was administered following a high-fat meal.
Period: Two-Sequence, Two-Way Crossover
Arm/Group | Diazepam Buccal Film, Then Diastat Rectal Gel | Diastat Rectal Gel, Then Diazepam Buccal Film | Diazepam Buccal Film Following a High-Fat Meal
Started | 15 | 16 | 0
Completed | 13 | 16 | 0
Not Completed | 2 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Period: DBF Following High-Fat Meal
Arm/Group | Diazepam Buccal Film, Then Diastat Rectal Gel | Diastat Rectal Gel, Then Diazepam Buccal Film | Diazepam Buccal Film Following a High-Fat Meal
Started | 0 (This arm did not continue in Period 2.) | 0 (This arm did not continue in Period 2.) | 10 (Participants in Period 2 completed 1 of the 2 arms in Period 1 and volunteered to continue.)
Completed | 0 | 0 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Enrolled participants in the study who received at least 1 dose of study medication.
Groups:
- Overall Population: 31 participants were enrolled and randomized to one of two treatment sequences with a 28-day washout period between doses:
  Treatment A was a single dose Diazepam Buccal Film administered on the inner aspect of the cheek according to the recommended dose regimen (10 mg to 17.5 mg according to body weight) following a moderate-fat meal.
  Treatment B was Diastat Rectal Gel administered rectally according to the package insert dosing instructions (10 mg to 20 mg according to body weight) following a moderate-fat meal.
  Treatment C was a voluntary second dose of Diazepam Buccal Film administered at the same dose and in the same manner as the earlier dose of Diazepam Buccal Film with the exception of administration following a high-fat meal.
Arm/Group | Overall Population
Number analyzed (Participants) | 31
Age, Continuous [Mean (Full Range); unit: years] | 40.4 [18 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: AUC 0-t
Description: Area Under Plasma Concentration-Time Curve From Time Zero to the last non-zero concentration
Time Frame: 0.5, 0.75, 1, 105, 2, 3, 4, 6, 9, 12, 24, 48, 72, 96, 120, 144, 192, and 240 hours post-dose
Population: Subjects who received both DBF and DRF administered following moderate fat meal with no significant violation of study restrictions, and for whom pharmacokinetic profile could be adequately characterized.
Measure: Geometric Mean (90% Confidence Interval); unit: hr*ng/mL
Groups:
- DBF Following Moderate-Fat Meal: Subjects received Diazepam Buccal Film administered on the inner aspect of the cheek following ingestion of a moderate-fat meal, allowing for transbuccal absorption of diazepam.
- DRG Following a Moderate Fat Meal: Subjects received Diastat AcuDial Rectal Gel administered rectally following ingestion of a moderate-fat meal, allowing for rectal absorption of diazepam.
- DBF Following a High Fat Meal: Subjects received Diazepam Buccal Film administered on the inner aspect of the cheek following ingestion of a high-fat meal, allowing for transbuccal absorption of diazepam.
Arm/Group | DBF Following Moderate-Fat Meal | DRG Following a Moderate Fat Meal | DBF Following a High Fat Meal
Number analyzed (Participants) | 29 | 28 | 10
hr*ng/mL | 7290.40 [5935.35 to 8954.81] | 5682.09 [4625.97 to 6979.31] | 8288.63 [6801.31 to 10100.00]

2. Primary Outcome: AUC 0-inf
Description: Area under concentration time curve, from time 0 extrapolated to infinity
Time Frame: 0.5, 0.75, 1, 105, 2, 3, 4, 6, 9, 12, 24, 48, 72, 96, 120, 144, 192, and 240 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (90% Confidence Interval); unit: hr*ng/mL
Groups:
- Diazepam Buccal Film Following a Moderate Fat Meal: Subjects received a single dose of Diazepam Buccal Film and Diastat Rectal Gel following a moderate-fat meal in a randomized sequence with a 28-day washout period between doses.
  Diazepam Buccal Film was administered on the inner aspect of the cheek according to the recommended dose regimen (10 mg to 17.5 mg according to body weight) allowing transbuccal absorption of diazepam.
- Diastat Rectal Gel Following a Moderate Fat Meal: Subjects received a single dose of Diazepam Buccal Film and Diastat Rectal Gel following a moderate-fat meal in a randomized sequence with a 28-day washout period between doses.
  Diastat Rectal Gel was administered rectally according to package insert dosing instructions (10 mg to 20 mg according to body weight) allowing rectal absorption of diazepam.
- Diazepam Buccal Film Following a High-Fat Meal: Subjects who volunteered to participate in the third period received a second dose of Diazepam Buccal Film in exactly the same manner as the earlier dose with the exception that the dose was administered following ingestion of a high-fat meal.
Arm/Group | Diazepam Buccal Film Following a Moderate Fat Meal | Diastat Rectal Gel Following a Moderate Fat Meal | Diazepam Buccal Film Following a High-Fat Meal
Number analyzed (Participants) | 29 | 27 | 10
hr*ng/mL | 8672.09 [7553.47 to 9956.32] | 6880.96 [5993.38 to 7899.98] | 8903.79 [7500.99 to 10568.93]

3. Primary Outcome: Cmax
Description: Maximum observed plasma concentration
Time Frame: 0.5, 0.75, 1, 105, 2, 3, 4, 6, 9, 12, 24, 48, 72, 96, 120, 144, 192, and 240 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (90% Confidence Interval); unit: ng/mL
Groups:
- Diazepam Buccal Film Following a Moderate-Fat Meal: Subjects received a single dose of Diazepam Buccal Film and Diastat Rectal Gel following a moderate-fat meal in a randomized sequence with a 28-day washout period between doses.
  Diazepam Buccal Film was administered on the inner aspect of the cheek according to the recommended dose regimen (10 mg to 17.5 mg according to body weight) allowing transbuccal absorption of diazepam.
- Diastat Rectal Gel Following a Moderate-Fat Meal: Subjects received a single dose of Diazepam Buccal Film and Diastat Rectal Gel following a moderate-fat meal in a randomized sequence with a 28-day washout period between doses.
  Diastat Rectal Gel was administered rectally according to package insert dosing instructions (10 mg to 20 mg according to body weight) allowing rectal absorption of diazepam.
Arm/Group | Diazepam Buccal Film Following a Moderate-Fat Meal | Diastat Rectal Gel Following a Moderate-Fat Meal | Diazepam Buccal Film Following a High-Fat Meal
Number analyzed (Participants) | 29 | 27 | 10
ng/mL | 204.25 [163.41 to 255.32] | 211.22 [168.98 to 264.02] | 181.61 [138.08 to 240.60]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time of signing the Informed Consent until at least 2 weeks following the last study drug administration (50 days overall).
Groups:
- Diazepam Buccal Film Following a Moderate-Fat Meal: Participants received a single dose of Diazepam Buccal Film and Diastat Rectal Gel following a moderate-fat meal in a randomized sequence with a 28-day washout period between doses.
  Diazepam Buccal Film was administered on the inner aspect of the cheek according to the recommended dose regimen (10 mg to 17.5 mg according to body weight) allowing transbuccal absorption of diazepam.
- Diastat Rectal Gel Following a Moderate-Fat Meal: Participants received a single dose of Diazepam Buccal Film and Diastat Rectal Gel following a moderate-fat meal in a randomized sequence with a 28-day washout period between doses.
  Diastat Rectal Gel was administered rectally according to package insert dosing instructions (10 mg to 20 mg according to body weight) allowing rectal absorption of diazepam.
- Diazepam Buccal Film Following a High-Fat Meal: Participants who volunteered to participate in the third period received a second dose of Diazepam Buccal Film in exactly the same manner as the earlier dose with the exception that the dose was administered following ingestion of a high-fat meal.
Arm/Group | Diazepam Buccal Film Following a Moderate-Fat Meal | Diastat Rectal Gel Following a Moderate-Fat Meal | Diazepam Buccal Film Following a High-Fat Meal
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/29 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/29 | 0/10
Other Adverse Events (participants affected / at risk) | 13/31 | 10/29 | 1/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diazepam Buccal Film Following a Moderate-Fat Meal (N=31) | Diastat Rectal Gel Following a Moderate-Fat Meal (N=29) | Diazepam Buccal Film Following a High-Fat Meal (N=10)
Somnolence (Nervous system disorders) | 7 (14) | 6 (14) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 2 (3) | 0 (0)
Sedation (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-05-24): https://cdn.clinicaltrials.gov/large-docs/20/NCT03953820/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-28): https://cdn.clinicaltrials.gov/large-docs/20/NCT03953820/SAP_001.pdf